CLINICAL TRIAL: NCT03388762
Title: A Randomized, Placebo-controlled Clinical Trial of a Polyherbal Dietary Supplement (GlucoSupreme™ Herbal) on Markers of Glycemic Control Among Prediabetic Adults
Brief Title: RCT of a Polyherbal Dietary Supplement for Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Alliance Institute for Integrative Medicine (Other)
Responsible Party: Principal Investigator, Chris D'Adamo, Director, Center for Integrative Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 022-DFH, HP-00075768
Record Dates: First submitted 2017-12-23; First posted 2018-01-03 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Prediabetic State
Keywords: Hyperglycemia; Prediabetes; Botanical; Phytochemicals; Dietary Supplements; Berberine; Fenugreek; American Ginseng; Gymnema; Banaba; Kudzu; Cinnamon; Glycated hemoglobin; Trigonella; Blood Glucose; Panax; Plant Extracts; Public Health; Chronic Disease
MeSH Terms: conditions — Prediabetic State; Hyperglycemia; Chronic Disease

STUDY DESIGN:
Intervention Model Description: This study is a 12-week, randomized, double-blinded, placebo-controlled clinical trial of GlucoSupreme™ Herbal. Eligible participants will be recruited from within participating clinical practices. All study outcomes will be biomarkers, capturing normal structure and function of the human body, derived from blood draws ordered during two physician visits spaced 12 weeks apart. This is a typical interval between blood assessments of glycemic control in routine clinical practice. An IRB-approved research associate will call each study participant at the 6-week mid-point of the study to assess compliance and collect data on any adverse events. Serious adverse events, while not anticipated, will be reported by the participant to a study physician as soon as possible.
Who Masked: Participant, Care Provider
Masking Description: The study products will be delivered to the investigative sites prior to enrollment of subjects. A study code will be provided for every batch of study product shipped to the investigational site prior to the beginning of the study. The placebo utilized in this clinical trial will be formulated to be as similar as possible to the active in appearance, odor, and other key characteristics, and packaging for both intervention and placebo will be the same. The de-identified study product will be packaged and labeled according to the study code and participant identification numbers; the Study Coordinator will oversee a locked master list of these, in addition to batch numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlucoSupreme™ Herbal (Active Comparator): Each daily serving of four GlucoSupreme™ Herbal tablets includes extracts from: cinnamon bark (Cinnamomum cassia) 500 mg, banaba leaf (Lagerstroemia speciosa standardized to 1% corosolic acid) 200 mg, kudzu root (Pueraria lobata standardized to 40% isoflavones) 200 mg, fenugreek seed (Trigonella foenum-graceum standardized to contain 60% saponins) 200 mg, and gymnema leaf (Gymnema sylvestre standardized to contain 25% gymnemic acid). Additionally, American ginseng root (Panax quinquefolius standardized to contain 5% ginsenosides) 200 mg, and berberine HCl derived from bark (Berberis aristata) 500 mg. Other ingredients include Cellulose (capsule), microcrystalline cellulose, silicon dioxide, and vegetable stearate.
  Interventions: Dietary Supplement: GlucoSupreme™ Herbal
- Control (Placebo Comparator): The placebo utilized in this clinical trial will be formulated by the manufacturer to be as similar as possible to the active intervention in appearance, odor, and other key characteristics. Packaging for the control will be identical to packaging for the Active Comparator.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: GlucoSupreme™ Herbal — This study will assess changes in glycemic parameters and other biomarkers over a twelve week period, with two blood draws (Baseline and 12 weeks). Additionally, an IRB-approved research associate will call each study participant at the 6-week mid-point of the study to assess compliance and collect data on any adverse events.
  Arms: GlucoSupreme™ Herbal
Other: Placebo — The placebo utilized in this clinical trial will be formulated by the manufacturer to be as similar as possible to the active intervention in appearance, odor, and other key characteristics. Packaging for the control will be identical to packaging for the Active Comparator.
  Arms: Control

SUMMARY:
The primary purpose of this study is to evaluate the impact of a polyherbal dietary supplement (Designs for Health - GlucoSupreme™ Herbal) on markers of glycemic control and other structure/function outcomes among a sample of prediabetic adults.

A 12-week randomized, double-blinded, placebo-controlled clinical trial will be conducted to achieve the purpose of this study. The research team hypothesizes that GlucoSupreme™ Herbal will improve a variety of validated markers of glycemic control that are commonly used in clinical practice more effectively than placebo.

DETAILED DESCRIPTION:
Prediabetes is a common state in which blood glucose levels are elevated, but are not elevated high enough to be considered Type 2 Diabetes (T2D). The worldwide prevalence of prediabetes is high and rapidly increasing. People with prediabetes are at increased risk for developing a variety of chronic diseases. Most notably, prediabetes nearly always precedes diagnosis of T2D, a poorly-controlled disease adversely affecting 14% of adults in the United States. T2D is responsible for increased risk of heart disease, stroke, blindness and other vision problems, kidney disease, amputations and death. Prediabetes often progresses to T2D relatively quickly, as pancreatic beta-cell dysfunction perpetuates. There are currently limited pharmacological options available for safely reducing the burden of prediabetes. Furthermore, these pharmacological options often carry potentially deleterious side effects. Low-risk alternatives are needed where lifestyle modifications, such as increased physical activity and weight loss, have failed.

Herbal dietary supplements have shown promise in safely managing impaired glycemic control in prediabetic adults in many clinical studies. A wide variety of herbs have been previously studied for these purposes, including cinnamon, fenugreek, banaba, curcumin, and a variety of combination products. Of these, most have demonstrated improved management of glycemic control, particularly with regard to reducing fasting blood glucose and postprandial glucose, HbA1c, fasting insulin levels, HOMA-Insulin Resistance, and increasing HOMA-β cell function among prediabetic adult populations. Many herbs have also demonstrated benefit in the management of glycemic control in clinical trials among T2D populations. These herbs include berberine, ginseng, gymnema, banaba, cinnamon, fenugreek, and kudzu, all of which are present in GlucoSupreme™ Herbal.

The research team hypothesizes that GlucoSupreme™ Herbal will demonstrate superior improvements in markers of glycemic control than placebo over twelve weeks of daily supplementation among a sample of healthy adults. The research team aims to conduct a randomized, placebo-controlled, double-blinded clinical trial to evaluate this hypothesis among a diverse sample of 40 prediabetic adults, and will implement a 1:1 study allocation ratio. This study will utilize an adaptive sample size re-estimation (SSR) approach where participant enrollment may be extended beyond the originally planned sample size if interim effect size is smaller than anticipated, but still promising, thereby preserving study power; this will be determined by examination of available unblinded endpoint data by an independent statistician after 30 subjects are enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Prediabetic blood measurement (HbA1C) of 5.7-6.4% and/or fasting blood glucose of 100-125 mg/dl and/or 2-hour Oral Glucose Tolerance Test blood glucose value of 140 mg/dl-199 mg/dl1 2) taken within the last 12 weeks
3. Agree to continue with current diet and refrain from taking any new nutritional or herbal supplements
4. Able to understand and write English
5. Voluntarily consent to the study and understand its nature and purpose including potential risks and side effects

Exclusion Criteria:

1. Current daily use of any oral hypoglycemic medication or insulin injection
2. Current daily use of any supplement containing the herbs in the study supplement
3. Known allergies to any substance in the study supplement
4. Current daily tobacco smoker
5. Currently pregnant or planning to become pregnant in the next 12 weeks
6. Any current or previous diagnosis of diabetes (Type 1 or Type 2)
7. Myocardial infarction, vascular surgery, or stroke in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Glucose | Baseline and study end (12 weeks from baseline)
  Elevated fasting blood glucose is one of the markers of the prediabetic state. According to American Diabetes Association criteria, the prediabetic fasting blood glucose range is 100 to 125 mg/dL (5.6 to 6.9 mmol/L). After fasting for 8-12 hours, > 0.5mL of blood will be collected from each participant, followed by centrifuge separation of plasma from cells within 45 minutes of collection. After maintaining the plasma fasting blood glucose at room temperature, it will be analyzed using standard enzymatic methodology.
Glycated hemoglobin/A1C (HbA1c) | Baseline and study end (12 weeks from baseline)
  Elevated HbA1c is another one of the markers of the prediabetic state and is defined as being within the range of 5.7-6.4%. A four mL sample of whole blood will be obtained from participants using techniques described above, and placed in an EDTA, lithium heparin, or sodium fluoride tube, followed by analysis using the Roche Tina Quant (Roche, Germany).
Fasting insulin | Baseline and study end (12 weeks from baseline)
  In prediabetes, pancreatic beta cells can no longer produce enough insulin to overcome insulin resistance, which can cause blood glucose levels to rise above the normal range. Thus, fasting insulin is a glycemic parameter of interest and is also used to determine insulin resistance. While normal values for fasting insulin are <25 microU/L, fasting insulin can vary widely among prediabetic individuals. After fasting for 8-12 hours, 0.8mL blood serum will be obtained from each participant. This fasting insulin assay will be performed using a 2-site electrochemiluminescent immunoassay on the Roche automated platform (Roche, Germany.).
Insulin Resistance (HOMA-IR) | Baseline and study end (12 weeks from baseline)
  Insulin resistance often sets the stage for progression to T2D by placing a high demand on insulin-producing beta cells during a prediabetic state. The advantage of using the validated HOMA-IR calculation is its relative simplicity and low-cost since it is derived from other primary outcomes of interest in this study. HOMA-IR is calculated as: [Fasting insulin (microU/L) x Fasting Blood Glucose (nmol/L)]/22.5.
β-cell function (HOMA-β) | Baseline and study end (12 weeks from baseline)
  Pancreatic beta cells (β-cells) produce insulin. Thus, their function is of interest in this prediabetic study population. As is the case with HOMA-IR, this formula utilizes values from our other study outcomes. HOMA- β is calculated as: (20 x Fasting insulin [microU/L])/(Fasting blood glucose [mmol/l] - 3.5).
Quantitative Insulin Sensitivity Check Index (QUICKI) | Baseline and study end (12 weeks from baseline)
  The validated QUICKI measurement to assess insulin sensitivity has also been studied in herbal dietary supplement clinical trials. QUICKI is calculated as: 1/(log-fasting blood glucose [mg/dL] + log-fasting insulin [uU/mL]).
Fructosamine | Baseline and study end (12 weeks from baseline)
  Many serum proteins are involved in glucose synthesis. Fructosamine represents the degree of glycation in these proteins, and is the concentration of plasma glucose over the lifetime of the protein. This useful test has been utilized in previous clinical studies of natural products3 4 and is an adjunct to the A1C and other fasting glycemic measurements, and reflects intermediate-term (previous 2-3 weeks) glycemic change. One mL of serum or plasma will be collected, followed by centrifuge separation within 45 minutes of collection, and analyzed using standard colorimetric assay methodology (LabCorp, Inc.).
GlycoMark | Baseline and study end (12 weeks from baseline)
  A blood test commonly used in clinical practice to determine peak hyperglycemia. The GlycoMark test provides accurate recognition of recent glycemic deterioration or improvement (within the previous 2-4 weeks)5 6 and is commonly given adjacently to A1C (a longer-term indicator of glycemic change) in clinical practice. One mL of serum or plasma will be collected, followed by centrifuge separation within 60 minutes of collection, and analyzed using standard enzymatic colorimetric assay methodology (LabCorp, Inc.).

SECONDARY OUTCOMES:
Lipid profile | Baseline and study end (12 weeks from baseline)
  A standard lipid panel consisting of total cholesterol, LDL, HDL, and triglycerides will be compared at baseline and the 12-week follow up visit. One mL of serum or plasma will be collected for all lipid parameters after 8 -12 hours of fasting and in the manner as described above, followed by centrifuge separation within 45 minutes of collection, and analyzed using standard enzymatic methodology (LabCorp, Inc.).
Inflammation | Baseline and study end (12 weeks from baseline)
  High-sensitivity C-reactive protein (Hs-CRP) is a common measure of inflammation that is commonly collected in clinical practice. Samples will undergo analysis by latex immunoturbidimetry on a COBAS Integra 800 (Roche, Germany).
Supplement compliance assessed using participant daily diary | Study end (12 weeks from baseline)
Adverse events | Throughout the study and at study end (12 weeks from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Chris D'Adamo, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - University of Maryland Center for Diabetes and Endocrinology, Baltimore, Maryland
  - University of Maryland Family Medicine Associates, Baltimore, Maryland
  - University of Maryland School of Medicine, Department of Family and Community Medicine, East Hall, Baltimore, Maryland
  - Alliance Integrative Medicine, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feinberg T, Wieland LS, Miller LE, Munir K, Pollin TI, Shuldiner AR, Amoils S, Gallagher L, Bahr-Robertson M, D'Adamo CR. Polyherbal dietary supplementation for prediabetic adults: study protocol for a randomized controlled trial. Trials. 2019 Jan 7;20(1):24. doi: 10.1186/s13063-018-3032-6. PMID 30616613